CLINICAL TRIAL: NCT04947774
Title: Real-world Study of Prophylactic Cranial Irradiation After Immunotherapy Combined With Chemotherapy for Extensive-stage Small Cell Lung Cancer
Brief Title: Prophylactic Cranial Irradiation in Extensive-stage Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Luhua Wang, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC2622
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Extensive-stage Small-cell Lung Cancer
Keywords: Small-cell Lung Cancer; Radiation:prophylactic cranial irradiation
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prophylactic cranial irradiation group: The extensive-stage SCLC patients will receive prophylactic cranial irradiation after standard first-line chemotherapy combined with immunotherapy, until disease progression or death.
  Interventions: Radiation: Prophylactic Cranial Irradiation
- Observation group: Patients with extensive-stage SCLC do not receive preventive craniocerebral irradiation after standard first-line chemotherapy combined with immunotherapy until the disease progresses or death.

INTERVENTIONS:
Radiation: Prophylactic Cranial Irradiation — The extensive-stage SCLC patients will receive prophylactic cranial irradiation ±immunotherapy after standard first-line chemotherapy combined with immunotherapy, until disease progression or death
  Other Names: Immunotherapy
  Groups: prophylactic cranial irradiation group

SUMMARY:
The prognosis of extensive-stage small cell lung cancer is still very poor, even for those who received chemotherapy and immunotherapy. This experimental study is a real-world research design to evaluate the effectiveness and safety of prophylactic cranial irradiation in patients with extensive-stage small cell lung cancer who with first-line chemotherapy combined with immunotherapy.

DETAILED DESCRIPTION:
This study is a prospective trial. This study included ES-SCLC patients who response after standard first-line treatment, and aimed to explore the safety and effectiveness of prophylactic cranial irradiation in this treatment modality.

The primary endpoint is progression-free survival in the brain.The secondary endpoints includes OS, PFS. The indicators for evaluating safety are the incidence and severity of adverse events.The exploratory endpoint is the molecular biomarkers for efficacy and toxicity predicting from tumor tissue and peripheral blood TMB.

The trial was designed by the National Cancer Center/Cancer Hospital of the Chinese Academy of Medical Sciences and Peking Union Medical College. The hypothesis is that preventive brain irradiation is safe and effective in the treatment of extensive SCLC combined with chemotherapy and immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent;
* With extensive small cell lung cancer;
* Previously received first-line standard chemotherapy, with treatment response of CR or PR;
* Can tolerate the radiotherapy process;
* Be over 18 years old
* Life expectancy ≥ 12 weeks;
* With the Eastern Cancer Cooperative Group (ECOG) score 0-1
* After the systemic treatment was received, there was no brain metastasis on MR before brain preventive irradiation.

Exclusion Criteria:

* Exclude subjects with central nervous system (CNS) metastasis at the first diagnosis;
* Pregnancy or breastfeeding;
* Any other conclusive medical, psychiatric and/or social reasons determined by the researcher;
* Subjects who have previously suffered from other malignant tumors (excluding non-melanoma skin cancer and the following carcinoma in situ: bladder, stomach, colon, endometrial, cervical/dysplasia, melanoma or breast cancer) are not allowed to participate in the study. Unless he/she has been in complete remission at least 2 years before enrolling in the study, and does not need to receive other treatments or does not need to receive other treatments during the study;
* Researchers believe that the treatment methods used in the study can cause harm or cause basic diseases whose toxicity is difficult to judge when judging adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to enroll patients who have completed and response to first-line chemotherapy combined with immunotherapy, Later immunotherapy treatments are open
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival in the brain | 1 year
  The length of time during and after treatment for a disease in which the patient lives with the disease but the intracranial lesions do not worsen

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  The length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse
Overall survival (OS) | 1 year
  The time from treatment to death from any cause
Adverse events | 1 year
  The incidence and severity of adverse events related to treatments
The cognitive function of the patient | 1 year
  Use the Montreal Cognitive Screening Scale (MoCA) to score, the total score is 30 points, ≥26 points are normal

OTHER OUTCOMES:
Exploratory end point including biomarkers | 1 year
  To explore the correlation of PD-L1 expression in tumor tissue , TCR, ctDNA in peripheral blood and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Bi Nan, MD, Study Director — Cancer Hospital, CAMS and PUMC
Locations (1):
- Cancer Insititute and Hosiptal of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Chen W, Zheng R, Zhang S, Zeng H, Zuo T, Xia C, Yang Z, He J. Cancer incidence and mortality in China in 2013: an analysis based on urbanization level. Chin J Cancer Res. 2017 Feb;29(1):1-10. doi: 10.21147/j.issn.1000-9604.2017.01.01. PMID 28373748
- [Background] Takada M, Fukuoka M, Kawahara M, Sugiura T, Yokoyama A, Yokota S, Nishiwaki Y, Watanabe K, Noda K, Tamura T, Fukuda H, Saijo N. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with cisplatin and etoposide for limited-stage small-cell lung cancer: results of the Japan Clinical Oncology Group Study 9104. J Clin Oncol. 2002 Jul 15;20(14):3054-60. doi: 10.1200/JCO.2002.12.071. PMID 12118018
- [Background] Halthore A, Goenka A, Sharma R, Knisely JPS. Prophylactic Cranial Irradiation for Resectable Small-Cell Lung Cancer. Clin Lung Cancer. 2018 Mar;19(2):115-119. doi: 10.1016/j.cllc.2017.08.004. Epub 2017 Aug 26. PMID 28958889
- [Background] Edelman MJ. Prophylactic Cranial Irradiation for Small-Cell Lung Cancer: Time for a Reassessment. Am Soc Clin Oncol Educ Book. 2020 May;40:24-28. doi: 10.1200/EDBK_281041. PMID 32421453
- [Background] Janne PA, Freidlin B, Saxman S, Johnson DH, Livingston RB, Shepherd FA, Johnson BE. Twenty-five years of clinical research for patients with limited-stage small cell lung carcinoma in North America. Cancer. 2002 Oct 1;95(7):1528-38. doi: 10.1002/cncr.10841. PMID 12237922
- [Background] Govindan R, Page N, Morgensztern D, Read W, Tierney R, Vlahiotis A, Spitznagel EL, Piccirillo J. Changing epidemiology of small-cell lung cancer in the United States over the last 30 years: analysis of the surveillance, epidemiologic, and end results database. J Clin Oncol. 2006 Oct 1;24(28):4539-44. doi: 10.1200/JCO.2005.04.4859. PMID 17008692
- [Background] Socinski MA, Smit EF, Lorigan P, Konduri K, Reck M, Szczesna A, Blakely J, Serwatowski P, Karaseva NA, Ciuleanu T, Jassem J, Dediu M, Hong S, Visseren-Grul C, Hanauske AR, Obasaju CK, Guba SC, Thatcher N. Phase III study of pemetrexed plus carboplatin compared with etoposide plus carboplatin in chemotherapy-naive patients with extensive-stage small-cell lung cancer. J Clin Oncol. 2009 Oct 1;27(28):4787-92. doi: 10.1200/JCO.2009.23.1548. Epub 2009 Aug 31. PMID 19720897
- [Background] Lara PN Jr, Natale R, Crowley J, Lenz HJ, Redman MW, Carleton JE, Jett J, Langer CJ, Kuebler JP, Dakhil SR, Chansky K, Gandara DR. Phase III trial of irinotecan/cisplatin compared with etoposide/cisplatin in extensive-stage small-cell lung cancer: clinical and pharmacogenomic results from SWOG S0124. J Clin Oncol. 2009 May 20;27(15):2530-5. doi: 10.1200/JCO.2008.20.1061. Epub 2009 Apr 6. PMID 19349543
- [Background] Rimner A, Wu AJ, Grills IS. What Is the Impact of Hippocampus Avoidance-Prophylactic Cranial Irradiation on Neurocognitive Preservation? J Thorac Oncol. 2021 May;16(5):722-724. doi: 10.1016/j.jtho.2021.02.026. No abstract available. PMID 33896571
- [Background] Wen P, Wang TF, Li M, Yu Y, Zhou YL, Wu CL. Meta-analysis of prophylactic cranial irradiation or not in treatment of extensive-stage small-cell lung cancer: The dilemma remains. Cancer Radiother. 2020 Feb;24(1):44-52. doi: 10.1016/j.canrad.2019.10.001. Epub 2020 Feb 7. PMID 32044160
- [Background] Spigel DR, Hainsworth JD, Shipley DL, Mekhail TM, Zubkus JD, Waterhouse DM, Daniel DB, Burris HA 3rd, Greco FA. Amrubicin and carboplatin with pegfilgrastim in patients with extensive stage small cell lung cancer: A phase II trial of the Sarah Cannon Oncology Research Consortium. Lung Cancer. 2018 Mar;117:38-43. doi: 10.1016/j.lungcan.2018.01.007. Epub 2018 Jan 12. PMID 29496254
- [Background] Pezzi TA, Fang P, Gjyshi O, Feng L, Liu S, Komaki R, Lin SH. Rates of Overall Survival and Intracranial Control in the Magnetic Resonance Imaging Era for Patients With Limited-Stage Small Cell Lung Cancer With and Without Prophylactic Cranial Irradiation. JAMA Netw Open. 2020 Apr 1;3(4):e201929. doi: 10.1001/jamanetworkopen.2020.1929. PMID 32236532
- [Background] Nosaki K, Seto T, Shimokawa M, Takahashi T, Yamamoto N. Is prophylactic cranial irradiation (PCI) needed in patients with extensive-stage small cell lung cancer showing complete response to first-line chemotherapy? Radiother Oncol. 2018 Jun;127(3):344-348. doi: 10.1016/j.radonc.2018.04.010. Epub 2018 May 7. PMID 29747871
- [Background] Yu J, Ouyang W, Yang Y, Zhang X, Zhou Y, Zhang J, Xie C. Prophylactic cranial irradiation for extensive-stage small cell lung cancer: Analysis based on active brain MRI surveillance. Clin Transl Radiat Oncol. 2020 Sep 15;25:16-21. doi: 10.1016/j.ctro.2020.09.005. eCollection 2020 Nov. PMID 32995574
- [Background] Ge W, Xu H, Yan Y, Cao D. The effects of prophylactic cranial irradiation versus control on survival of patients with extensive-stage small-cell lung cancer: a meta-analysis of 14 trials. Radiat Oncol. 2018 Aug 23;13(1):155. doi: 10.1186/s13014-018-1101-3. PMID 30139360